CLINICAL TRIAL: NCT02016534
Title: A Multicenter, Phase 2, Single Arm, Two Cohort Study Evaluating the Efficacy, Safety, and Pharmacokinetics of AMG337 in Subjects With MET Amplified Gastric/Gastroesophageal Junction/Esophageal Adenocarcinoma or Other MET Amplified Solid Tumors
Brief Title: Phase 2 Study of AMG 337 in MET Amplified Gastric/Esophageal Adenocarcinoma or Other Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Amgen decision following interim review of efficacy and safety data from the AMG 337 program.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130111; 2013-001277-24 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Stomach Neoplasms
Keywords: MET Amplified Gastric / Gastroesophageal Junction / Esophageal Adenocarcinoma, or other solid tumors.
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — AMG 337

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): AMG 337 Monotherapy
  Interventions: Drug: AMG 337

INTERVENTIONS:
Drug: AMG 337 — AMG 337 300mg orally daily.

SUMMARY:
This is a multi-centre Phase 2 study. The study will evaluate the activity and safety of AMG 337 in patients who have MET amplified gastric, gastroesophageal junction or esophageal adenocarcinoma or other MET amplified solid tumors. The study is designed to estimate the objective response rate of AMG 337 by tumor type.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, single arm, 2 cohort study to assess the safety, efficacy and pharmacokinetics of AMG 337 in MET amplified Gastric/esophageal adenocarcinoma or other solid tumors. Approximately 140 subjects will be enrolled to either Cohort 1 (subjects with MET amplified G/E adenocarcinoma with measurable tumor) or Cohort 2 (subjects with MET amplified solid tumors with measurable tumor/up to 10 subjects with MET amplified G/E adenocarcinoma with non-measurable tumor/up to 10 subjects who have received prior MET antibody therapy). All subjects will self-administer AMG 337 300 mg daily until disease progression or other protocol specified end of treatment criteria is met.

Tumor tissue, biomarkers, Pharmacokinetics and Patient reported Outcomes will all be assessed.

Tumor assessment by RECIST 1.1 will be followed during study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to daily self-administer AMG 337 orally as a whole capsule
* Male or female 18 years of age or over.
* Pathologically confirmed advanced G/GEJ/E adenocarcinoma (Cohort 1) or other solid tumor (Cohort 2) for which subject has received prior therapy for advanced disease, for which no standard therapy exists, or subject refuses standard therapy
* Tumor MET amplified by protocol-specified centralized testing.
* Measurable disease per RECIST 1.1 guidelines. Cohort 2 may include up to 10 subjects with advanced MET amplified, G/GEJ/E adenocarcinoma with non-measurable tumor per RECIST v1.1
* (ECOG) Performance Status of 0, 1 or 2

Exclusion Criteria:

* Known central nervous system metastases
* Candidate for curative surgery or definitive chemoradiation
* Peripheral edema > grade 1
* Persistent gastric outlet obstruction, complete dysphagia or are dependent upon jejunostomy for feeding. Significant gastrointestinal disorder(s) that in the opinion of the Investigator may influence drug absorption
* Acute Hepatitis B. Chronic Hepatitis B eligible if condition is stable and, in the opinion of the investigator or Amgen physician, if consulted, would not pose a risk to subject safety
* Detectable Hepatitis C virus (indicative of active Hepatitis C)
* Currently receiving any anti-tumor treatments, or less than 14 days prior to enrollment since ending anti-tumor treatment
* Prior treatment with small molecule inhibitors of the MET pathway.

Other protocol defined inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (RECIST v1.1) in subjects with MET Amplified measurable G/GEJ/E adenocarcinoma (Cohort 1) | 2.5 years
  Determine antitumor activity of AMG 337 in subjects with MET amplified G/GEJ/E adenocarcinoma

SECONDARY OUTCOMES:
Duration of response (cohort 1 and subjects with measurable disease at baseline in cohort 2) | 2.5 years
Time to response (Cohort 1 and subjects with measurable disease at baseline in cohort 2) | 2.5 years
Progression free survival | 2.5 years
Overall survival | 2.5 years
Incidence and severity of adverse events and significant laboratory abnormalities | 2.5 years
AMG 337 exposure and dose intensity | 2.5 years
Pharmacokinetic parameters | 2.5 years
  Including, but not limited to, minimum (trough) concentrations at pre-dose times, maximum concentrations (C max), the time of C max (t max), and area under the plasma concentration - time curve (AUC).
Objective Response Rate (per RECIST v1.1) in subjects with other MET amplified solid tumors (subjects with measurable disease in cohort 2). | 2.5 years
  Determine antitumor activity of AMG 337 in subjects with other MET amplified solid tumors.

OTHER OUTCOMES:
Patient Reported Outcomes (PRO) Health related quality of life (HRQoL) | 3 years
  To evaluate the impact of AMG 337 on health-related quality of life (HRQoL) in subjects with MET amplified G/GEJ/E adenocarcinoma (Cohort 1 only).
Tumor tissue and circulating serum biomarkers | 3 years
  assessed at baseline. Circulating tumor cells (CTC) and circulating serum biomarkers will also be assessed at baseline and during study treatment
Prediction of response rates to AMG 337 by analysing tumor DNA for MET pathway-related genes | 3 years
  To analyse tumor DNA samples for MET pathway-related genes (and other genes based on emerging data) that may predict response to AMG 337
Response to AMG 337 and MET amplification, expression or presence of mutation in tumor specimens | 3 years
  Explore whether the level of MET amplification, expression, or presence of mutation in tumor specimens correlates with response to AMG 337.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (81):
- United States (6):
  - Research Site, New Haven, Connecticut
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Seattle, Washington
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Kurralta Park, South Australia
  - Research Site, Bentleigh East, Victoria
  - Research Site, Heidelberg, Victoria
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Wels
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Research Site, Edmonton, Alberta, Canada
- Research Site, Santiago, Chile
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (8):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Reims
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Germany (4):
  - Research Site, Cologne
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, München
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion - Crete
  - Research Site, Ioannina
  - Research Site, Piraeus
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Szolnok
- Italy (14):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cremona
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano MI
  - Research Site, Torino
  - Research Site, Udine
- Research Site, Lima, Peru
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Konin
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (3):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Hwasun
  - Research Site, Seoul
- Spain (4):
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid
- United Kingdom (6):
  - Research Site, Edinburgh
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Sutton

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com